CLINICAL TRIAL: NCT02038452
Title: Randomised, Multicentre, Open Label, Parallel Group Pragmatic Clinical Trial of Local Steroid Injection Versus Night Splinting in Mild to Moderate Carpal Tunnel Syndrome (CTS)
Brief Title: Injection Versus Splinting in Carpal Tunnel Syndrome
Acronym: INSTinCTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keele University (Other)
Collaborators: Arthritis Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 464/11; 20105 (Other Grant/Funding Number: Arthritis Research UK); 2013-001435-48 (EudraCT Number); 13/NW/0280 (Other: UK NHS Research Ethics Committee); 09392969 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2014-01-09; First posted 2014-01-16 (Estimated); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: hand; wrist; carpal; tunnel; syndrome; pragmatic; randomised; steroid; splint
MeSH Terms: conditions — Carpal Tunnel Syndrome; Syndrome | interventions — Methylprednisolone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroid Injection (Active Comparator): Single steroid injection into Carpal Tunnel (as Depo-medrone 20mg)
  Interventions: Drug: Depo-Medrone
- Wrist Splint (Active Comparator): Wrist splint to be worn at night
  Interventions: Device: Wrist Splint

INTERVENTIONS:
Drug: Depo-Medrone — Steroid Injection
  Arms: Steroid Injection
Device: Wrist Splint — Simple wrist splint
  Other Names: Generic wrist splint
  Arms: Wrist Splint

SUMMARY:
Carpal Tunnel Syndrome (CTS) is a common condition in which a nerve (known as the median nerve) is squeezed where it passes through the wrist. It can cause pain or aching, tingling or numbness in the affected hand. It may disturb sleep, or affect ability to do day to day things.

There have been several studies into the best treatment of patients with severe symptoms of CTS who are referred to a hospital for treatment. However, little is known about the best treatments for patients with mild to moderate symptoms who visit their GP but do not require hospital treatment.

The study will investigate whether a steroid injection is clinically effective in reducing symptoms and improving function in the short term (6 weeks) compared to a night splint in people consulting with mild to moderate CTS in primary care.We will study the effects of these 2 treatments over 6 weeks and at 6 months. Subject to further funding, the Study will also look at whether these 6 weeks of treatment are effective 1 year and 2 years later.

The study will take place in up to 50 GP practices and hospital clinics across the UK. Patients aged 18 and over who have been diagnosed with mild to moderate CTS which has been present for at least 6 weeks will be eligible for inclusion.

The steroid is a drug called "DepoMedrone." This drug is already widely used to treat CTS. In this study, one injection will be given. The splint is made of elastic and has an aluminium bar which sits on the palm of the hand. In this study, the splint will be worn at night for 6 weeks. Each participant will receive either a single steroid injection or a splint, and will be asked to complete up to 5 questionnaires over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* A clinical diagnosis of unilateral or bilateral CTS as made by a GP or trained clinician according to the diagnostic criteria
* Mild (e.g. intermittent paraesthesia) or moderate (e.g. constant paraesthesia, reversible numbness and / or pain) severity CTS of idiopathic nature
* Symptom duration of episode of at least 6 weeks
* Written informed consent provided by the patient, prior to any trial specific procedures

Exclusion Criteria:

* Steroid injection or night splints for CTS in the affected wrist within preceding 6 months
* Any previous surgery on the affected wrist
* Severe CTS exhibiting constant numbness or pain, constant sensory loss, severe thenar muscle atrophy or symptom severity which requires the patient to be referred for a surgical opinion
* Clinical suspicion of local or systemic sepsis or infection
* Current or previous infection of the affected wrist
* Trauma to the affected hand requiring surgery or immobilisation in the previous 12 months
* Unable to tolerate the study interventions
* Unable to understand and complete self-report questionnaires written in English
* Inter-current illness including, but not limited to:

  * poorly controlled thyroid disease
  * poorly controlled diabetes mellitus
  * vibration-induced neuropathy
  * inflammatory joint disease
  * suspected complex neurological conditions
  * any other severe medical illness which in the opinion of the local Principal Investigator (or other authorised clinical delegate) precludes trial participation
* Pregnant or lactating females
* Receiving anticoagulants
* Any history of hypersensitivity to Depo-Medrone or any of its excipients
* Allergy to any of the splint materials
* Known abuse of drugs or alcohol
* Involved in on-going litigation cases for their condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12-31 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Roddy, Fellow RCP, Principal Investigator — Keele University
Locations (1):
- Staffordshire and Stoke on Trent Partnership NHS Trust, Newcastle-under-Lyme, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Keele University is a member of the UK Reproducibility Network and committed to the principles of the UK Concordat on Open Research Data. The School of Medicine and Keele Clinical Trials Unit have a longstanding commitment to sharing data from our studies to improve research reproducibility and to maximise benefits for patients, the wider public, and the health and care system. We encourage collaboration with those who collected the data, to recognise and credit their contributions.
  The School of Medicine and Keele Clinical Trials Unit make data available to bona-fide researchers upon reasonable request via open or restricted access through a strict controlled access procedure. The release of data may be subject to a data use agreement (DUA) between the Sponsor and the third party requesting the data. In the first instance, data requests and enquiries should be directed to medicine.datasharing@keele.ac.uk.

REFERENCES:
- [Background] Chesterton LS, Dziedzic KS, van der Windt DA, Davenport G, Myers HL, Rathod T, Blagojevic-Bucknall M, Jowet SM, Burton C, Roddy E, Hay EM. The clinical and cost effectiveness of steroid injection compared with night splints for carpal tunnel syndrome: the INSTINCTS randomised clinical trial study protocol. BMC Musculoskelet Disord. 2016 Oct 6;17(1):415. doi: 10.1186/s12891-016-1264-8. PMID 27716159
- [Result] Chesterton LS, Blagojevic-Bucknall M, Burton C, Dziedzic KS, Davenport G, Jowett SM, Myers HL, Oppong R, Rathod-Mistry T, van der Windt DA, Hay EM, Roddy E. The clinical and cost-effectiveness of corticosteroid injection versus night splints for carpal tunnel syndrome (INSTINCTS trial): an open-label, parallel group, randomised controlled trial. Lancet. 2018 Oct 20;392(10156):1423-1433. doi: 10.1016/S0140-6736(18)31572-1. PMID 30343858

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 25 General Practices and community musculoskeletal clinics between 17/04/2014 and 31/12/2016.
Pre-assignment Details: Patients with a positive carpal tunnel syndrome (CTS) diagnosis were assessed for eligibility by the GP/clinician based on the inclusion/exclusion criteria. Patients who were interested in trial participation were then seen by appropriate member of the clinical team who explained the trial in full, and were asked to provide written informed consent.
  750 patients were assessed for eligibility. 405 were eligible and 234 subsequently consented to randomisation.
Period: Overall Study
Arm/Group | Steroid Injection | Wrist Splint
Started | 116 | 118
Baseline | 113 | 117
6 Weeks Follow-up | 108 | 109
6 Months Follow-up | 96 | 97
12 Months Follow-up | 87 | 88
24 Months Follow-up | 78 | 81
Completed | 78 | 81
Not Completed | 38 | 37
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Lost to Follow-up | 31 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid Injection | Wrist Splint | Total
Number analyzed (Participants) | 116 | 118 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (17.0) | 52.2 (14.9) | 52.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 81 | 154
  Male | 43 | 37 | 80
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 116 | 118 | 234
First time diagnosed with carpal tunnel syndrome [Count of Participants; unit: Participants]
  Yes | 97 | 102 | 199
  No | 16 | 15 | 31
  Missing | 3 | 1 | 4
Number of times previously had carpal tunnel syndrome [Count of Participants; unit: Participants]
  N/A | 97 | 102 | 199
  1 | 11 | 8 | 19
  2 | 1 | 1 | 2
  3 | 0 | 0 | 0
  More than 3 | 3 | 4 | 7
  Missing | 4 | 3 | 7
Hand or wrist previously affected by carpal tunnel syndrome [Count of Participants; unit: Participants]
  N/A | 97 | 102 | 199
  Right | 6 | 3 | 9
  Left | 1 | 2 | 3
  Both | 8 | 9 | 17
  Missing | 4 | 2 | 6
Treatment for previous carpal tunnel syndrome [Number; unit: participants] — Participants may select more than one treatment.
  participants
    N/A | 97 | 102 | 199
    Steroid injection | 3 | 4 | 7
    Wrist splint | 7 | 4 | 11
    Carpal tunnel decompression | 3 | 2 | 5
    Ultrasound | 1 | 1 | 2
    Exercises | 0 | 0 | 0
    Vitamin supplements | 0 | 1 | 1
    Changes in workplace | 0 | 0 | 0
    Other | 1 | 0 | 1
    None | 5 | 8 | 13
Steroid injection into a joint other than wrist if previously had carpal tunnel syndrome [Count of Participants; unit: Participants]
  N/A | 97 | 102 | 199
  Yes | 9 | 9 | 18
  No | 7 | 6 | 13
  Missing | 3 | 1 | 4
Usefulness of injection into other joint if previously had carpal tunnel syndrome [Count of Participants; unit: Participants]
  N/A | 104 | 108 | 212
  Of great help | 7 | 7 | 14
  Of some help | 1 | 1 | 2
  Of little help | 0 | 0 | 0
  Of no help | 1 | 1 | 2
  Missing | 3 | 1 | 4
Which problematic hand or wrist [Count of Participants; unit: Participants]
  Right | 36 | 37 | 73
  Left | 19 | 20 | 39
  Both | 57 | 59 | 116
  Missing | 4 | 2 | 6
If both hands problematic, which hand was worse [Count of Participants; unit: Participants]
  N/A | 55 | 57 | 112
  Right | 25 | 24 | 49
  Left | 13 | 19 | 32
  No difference | 7 | 3 | 10
  Missing | 16 | 15 | 31
Dominant hand [Count of Participants; unit: Participants]
  Right | 99 | 99 | 198
  Left | 12 | 16 | 28
  Missing | 5 | 3 | 8
Duration of hand or wrist problems [Count of Participants; unit: Participants]
  <3 months | 19 | 17 | 36
  3-6 months | 37 | 33 | 70
  6 months-1 year | 22 | 27 | 49
  >1 year | 34 | 39 | 73
  Missing | 4 | 2 | 6
How did your hand or wrist problems start [Count of Participants; unit: Participants]
  Suddenly | 33 | 17 | 50
  Gradually | 79 | 99 | 178
  Missing | 4 | 2 | 6
Particular position causes hand or wrist problems [Count of Participants; unit: Participants]
  Yes | 50 | 62 | 112
  No | 62 | 54 | 116
  Missing | 4 | 2 | 6
Curently taking pain relief [Count of Participants; unit: Participants]
  Yes | 36 | 34 | 70
  No | 77 | 83 | 160
  Missing | 3 | 1 | 4
Number of times a day taking pain relief [Count of Participants; unit: Participants]
  N/A | 77 | 83 | 160
  1 | 7 | 8 | 15
  2 | 13 | 5 | 18
  3 | 5 | 5 | 10
  4 | 3 | 5 | 8
  5 | 0 | 1 | 1
  Missing | 11 | 11 | 22
Number of days per week taking pain relief [Count of Participants; unit: Participants]
  N/A | 77 | 83 | 160
  1 | 0 | 0 | 0
  2 | 1 | 4 | 5
  3 | 3 | 0 | 3
  4 | 1 | 0 | 1
  5 | 2 | 2 | 4
  6 | 0 | 0 | 0
  7 | 14 | 7 | 21
  Missing | 18 | 22 | 40
Number of weeks in a month taking pain relief [Count of Participants; unit: Participants]
  N/A | 77 | 83 | 160
  1 | 1 | 0 | 1
  2 | 2 | 1 | 3
  3 | 1 | 0 | 1
  4 | 17 | 9 | 26
  Missing | 18 | 25 | 43
In a current paid job [Count of Participants; unit: Participants]
  Yes | 58 | 74 | 132
  No | 55 | 42 | 97
  Missing | 3 | 2 | 5
If not in a current paid job, describe current position [Number; unit: participants] — Participants may select more than one option
  participants
    N/A | 58 | 74 | 132
    Retired | 38 | 29 | 67
    Student | 3 | 1 | 4
    Looking after children/home | 12 | 9 | 21
    Unemployed | 3 | 7 | 10
    Voluntary worker | 2 | 0 | 2
Typical weekly working hours [Count of Participants; unit: Participants]
  N/A | 55 | 42 | 97
  Full time | 39 | 47 | 86
  Part time | 18 | 27 | 45
  Missing | 4 | 2 | 6
Describes current situation in respect of your job [Count of Participants; unit: Participants]
  N/A | 55 | 42 | 97
  Doing my usual job | 50 | 62 | 112
  On paid annual leave/holiday | 2 | 1 | 3
  Working fewer hours | 1 | 2 | 3
  Doing lighter duties | 1 | 6 | 7
  On paid sick leave | 3 | 3 | 6
  On unpaid sick leave | 0 | 0 | 0
  Missing | 4 | 2 | 6
If not doing usual job/annual leave, is this due to your hand or wrist problems [Count of Participants; unit: Participants]
  N/A | 105 | 105 | 210
  Yes | 2 | 4 | 6
  No | 3 | 6 | 9
  Missing | 6 | 3 | 9
Taken time off work during the last 6 months for your hand or wrist problems [Count of Participants; unit: Participants]
  N/A | 55 | 42 | 97
  Yes | 8 | 5 | 13
  No | 49 | 69 | 118
  Missing | 4 | 2 | 6
I feel my welfare is important to my employer [Count of Participants; unit: Participants]
  N/A | 104 | 111 | 215
  Strongly disagree | 0 | 0 | 0
  Disagree | 0 | 0 | 0
  Agree | 4 | 3 | 7
  Strongly agree | 4 | 2 | 6
  Missing | 4 | 2 | 6
Which treatment would you prefer [Count of Participants; unit: Participants]
  Strongly prefer wrist injection | 13 | 13 | 26
  Somewhat prefer wrist injection | 11 | 21 | 32
  No preference | 65 | 60 | 125
  Somewhat prefer night splints | 12 | 8 | 20
  Strongly prefer night splints | 6 | 10 | 16
  Missing | 9 | 6 | 15
If you had received wrist injection, would you expect your symptoms to improve [Count of Participants; unit: Participants]
  Yes | 69 | 70 | 139
  No | 0 | 2 | 2
  Not sure | 39 | 41 | 80
  Missing | 8 | 5 | 13
If you received night splint, would you expect your symptoms to improve [Count of Participants; unit: Participants]
  Yes | 46 | 40 | 86
  No | 3 | 4 | 7
  Not sure | 58 | 69 | 127
  Missing | 9 | 5 | 14
My hand or wrist problem will last for a long time [Count of Participants; unit: Participants]
  Strongly disagree | 3 | 3 | 6
  Disagree | 7 | 8 | 15
  Neither agree nor disagree | 45 | 51 | 96
  Agree | 44 | 42 | 86
  Strongly agree | 14 | 12 | 26
  Missing | 3 | 2 | 5
My hand or wrist problem has major consequences on my life [Count of Participants; unit: Participants]
  Strongly disagree | 4 | 10 | 14
  Disagree | 19 | 22 | 41
  Neither agree nor disagree | 26 | 30 | 56
  Agree | 41 | 37 | 78
  Strongly agree | 23 | 17 | 40
  Missing | 3 | 2 | 5
There is a lot that I can do to control my hand or wrist problems [Count of Participants; unit: Participants]
  Strongly disagree | 12 | 9 | 21
  Disagree | 21 | 31 | 52
  Neither agree nor disagree | 48 | 42 | 90
  Agree | 30 | 32 | 62
  Strongly agree | 2 | 2 | 4
  Missing | 3 | 2 | 5
What I can do determines whether my hand or wrist problems gets better or worse [Count of Participants; unit: Participants]
  Strongly disagree | 4 | 4 | 8
  Disagree | 11 | 14 | 25
  Neither agree nor disagree | 40 | 32 | 72
  Agree | 49 | 57 | 106
  Strongly agree | 9 | 9 | 18
  Missing | 3 | 2 | 5
Treatment can control my hand or wrist problem [Count of Participants; unit: Participants]
  Strongly disagree | 0 | 0 | 0
  Disagree | 3 | 0 | 3
  Neither agree nor disagree | 20 | 35 | 55
  Agree | 74 | 71 | 145
  Strongly agree | 16 | 9 | 25
  Missing | 3 | 3 | 6
My hand or wrist problem affects me emotionally [Count of Participants; unit: Participants]
  Strongly disagree | 10 | 18 | 28
  Disagree | 17 | 19 | 36
  Neither agree nor disagree | 17 | 21 | 38
  Agree | 40 | 45 | 85
  Strongly agree | 29 | 13 | 42
  Missing | 3 | 2 | 5
Been bother by feeling down, depressed or hopeless [Count of Participants; unit: Participants]
  Yes | 47 | 39 | 86
  No | 66 | 78 | 144
  Missing | 3 | 1 | 4
Been bothered by little interest or pleasure in doing things [Count of Participants; unit: Participants]
  Yes | 39 | 33 | 72
  No | 74 | 83 | 157
  Missing | 3 | 2 | 5
Diagnosed with hypothyroidism [Count of Participants; unit: Participants]
  Yes | 5 | 9 | 14
  No | 108 | 107 | 215
  Missing | 3 | 2 | 5
Diagnosed with diabetes [Count of Participants; unit: Participants]
  Yes | 13 | 8 | 21
  No | 99 | 109 | 208
  Missing | 4 | 1 | 5
Any other conditions affecting neck, shoulders or elbows [Count of Participants; unit: Participants]
  Yes | 45 | 28 | 73
  No | 68 | 88 | 156
  Missing | 3 | 2 | 5
Had pain anywhere else [Count of Participants; unit: Participants]
  Yes | 74 | 72 | 146
  No | 39 | 45 | 84
  Missing | 3 | 1 | 4
Last time you were free of pain [Count of Participants; unit: Participants]
  <3 months ago | 22 | 20 | 42
  3-6 months ago | 13 | 19 | 32
  6 months-1 year ago | 9 | 23 | 32
  1-3 years ago | 38 | 23 | 61
  >3 years ago | 31 | 32 | 63
  Missing | 3 | 1 | 4
On average, how often do you drink alcohol [Count of Participants; unit: Participants]
  Daily or most days | 11 | 11 | 22
  Once or twice a week | 38 | 45 | 83
  Once or twice a month | 25 | 22 | 47
  Once or twice a year | 16 | 18 | 34
  Never | 23 | 21 | 44
  Missing | 3 | 1 | 4
What is your current smoking status [Count of Participants; unit: Participants]
  Never smoked | 55 | 55 | 110
  Previously smoked | 39 | 48 | 87
  Current smoker | 19 | 13 | 32
  Missing | 3 | 2 | 5
Has insomnia due to hand or wrist problem [Count of Participants; unit: Participants] — Participants were asked four questions how hand and wrist problems affects their sleep. Participants reporting hand and wrist problems affects their sleep on most nights on one or more questions were deemed to have insomnia. Based on multiply imputed data.
  Participants
    No | 46 | 58 | 104
    Yes | 70 | 60 | 130
To what extent have hand or wrist problems affected your performance at work over the past month [Mean (Standard Deviation); unit: units on a scale] — 0-10 scale; 0=not at all, 10=unable to do job
  units on a scale | 3.8 (3.0) | 4.2 (2.9) | 4.0 (3.0)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 30.2 (7.6) | 30.5 (7.5) | 30.4 (7.6)
Boston carpal tunnel symptom severity and functional limitations [Mean (Standard Deviation); unit: units on a scale] — Scale 1-5, higher scores indicate more symptom severity and functional limitations. Analysis is based on multiply imputed data.
  units on a scale | 2.69 (0.70) | 2.65 (0.62) | 2.67 (0.66)
Boston carpal tunnel symptom severity subscale [Mean (Standard Deviation); unit: units on a scale] — Scale 1-5, higher scores indicate more severe symptoms. Analysis is based on multiply imputed data.
  units on a scale | 2.96 (0.66) | 2.91 (0.61) | 2.94 (0.63)
Boston carpal tunnel functional limitations subscale [Mean (Standard Deviation); unit: units on a scale] — Scale 1-5, higher scores indicate more severe functional impairment. Analysis is based on multiply imputed data.
  units on a scale | 2.32 (0.92) | 2.28 (0.84) | 2.30 (0.88)
Hand-wrist pain intensity [Mean (Standard Deviation); unit: units on a scale] — 0-10 scale, higher scores indicating more pain. Analysis is based on multiply imputed data.
  units on a scale | 6.33 (2.05) | 6.12 (2.21) | 6.23 (2.13)

OUTCOME MEASURES:

1. Primary Outcome: Symptom Severity and Limitations in Hand Function as Assessed by the BCTQ 6 Weeks
Description: Comparison of overall BCTQ between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms and functional impairment). BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
score on a scale | 2.02 (0.81) | 2.29 (0.75)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p < 0.001, Regression, Linear; Multiple imputation for missing data was performed. Linear regression adjusted for baseline score, sex, age, and duration of symptoms; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.48 to -0.16]

2. Secondary Outcome: BCTQ Symptom Severity Subscale 6 Weeks
Description: Comparison of BCTQ symptom severity between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms). BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
score on a scale | 2.12 (0.84) | 2.43 (0.76)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p < 0.001, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.53 to -0.17]

3. Secondary Outcome: BCTQ Functional Limitations Subscale 6 Weeks
Description: Comparison of BCTQ functional limitations between treatment groups at 6 weeks follow-up (1-5 scale, higher score indicates more severe functional impairment). BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
score on a scale | 1.88 (0.88) | 2.09 (0.86)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.003, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.43 to -0.09]

4. Secondary Outcome: Hand-wrist Pain Intensity 6 Weeks
Description: Comparison of pain scores between treatment groups at 6 weeks follow-up (0-10 scale, higher score indicates more pain).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
units on a scale | 3.42 (2.77) | 4.28 (2.73)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.005, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.64 to -0.30]

5. Secondary Outcome: Insomnia Due to Hand-wrist Problems 6 Weeks
Description: Participants were asked four questions how hand and wrist problems affects their sleep. Participants reporting hand and wrist problems affects their sleep on most nights on one or more questions were deemed to have insomnia.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
Participants
  No | 83 | 73
  Yes | 33 | 45
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.018, Regression, Logistic; Multiple imputation for missing data was performed. Logistic regression adjusted for baseline score, sex, age, and duration of symptoms; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.22 to 0.87]

6. Secondary Outcome: Referral for Surgery 6 Weeks
Description: Participants were asked if they were referred for surgery (carpal tunnel decompression) in the last 6 weeks. Multiple imputation for missing data was performed at 6 weeks. Comparison of outcome between treatment arms planned to adjust for sex, age, and duration of symptoms. Logistic regression was not performed due to small number of 'yes' counts.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
Participants
  No | 112 | 113
  Yes | 4 | 5

7. Secondary Outcome: Surgery 6 Weeks
Description: Participants were asked if they had surgery for carpal tunnel syndrome in the last 6 weeks. Multiple imputation for missing data was performed at 6 weeks. Comparison of outcome between treatment arms planned to adjust for sex, age, and duration of symptoms. Logistic regression was not performed due to small number of 'yes' counts.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
Participants
  No | 114 | 116
  Yes | 2 | 2

8. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Months
Description: Comparison of overall BCTQ between treatment groups at 6 months follow-up (1-5 scale, higher score indicates more severe symptoms and functional impairment). BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
score on a scale | 2.15 (0.79) | 2.06 (0.73)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.500, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.11 to 0.23]

9. Secondary Outcome: BCTQ Symptom Severity Subscale 6 Months
Description: Comparison of BCTQ symptom severity between treatment groups at 6 months follow-up (1-5 scale, higher score indicates more severe symptoms). BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
score on a scale | 2.33 (0.86) | 2.18 (0.75)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.21, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.07 to 0.33]

10. Secondary Outcome: BCTQ Functional Limitations Subscale 6 Months
Description: Comparison of BCTQ functional limitations between treatment groups at 6 months follow-up (1-5 scale, higher score indicates more functional impairment). BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
score on a scale | 1.91 (0.84) | 1.89 (0.84)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.96, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.175 to 0.166]

11. Secondary Outcome: Hand-wrist Pain Intensity 6 Months
Description: Comparison of pain scores between treatment groups at 6 months follow-up. 0-10 scale, higher score indicates more pain.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
units on a scale | 4.32 (3.26) | 3.46 (3.01)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.055, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.02 to 1.59]

12. Secondary Outcome: Insomnia Due to Hand-wrist Problems 6 Months
Description: as for outcome 5
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
Participants
  No | 79 | 86
  Yes | 37 | 32
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.76, Regression, Logistic; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.55 to 2.20]

13. Secondary Outcome: Referral to Surgery 6 Months
Description: Participants were asked if they were referred for surgery (carpal tunnel decompression) in the last 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
Participants
  No | 94 | 104
  Yes | 22 | 14
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.23, Regression, Logistic; Multiple imputation for missing data was performed. Logistic regression for sex, age, and duration of symptoms; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.73 to 3.77]

14. Secondary Outcome: Surgery 6 Months
Description: Participants were asked if they had surgery for carpal tunnel syndrome in the last 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
Participants
  No | 99 | 105
  Yes | 17 | 13
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.66, Regression, Logistic; Multiple imputation for missing data was performed. Logistic regression adjusted for sex, age, and duration of symptoms; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.41 to 3.98]

15. Secondary Outcome: Herbal Remedies and Vitamin Use 6 Months
Description: Participants were asked if they had bought herbal remedies or vitamins to help with hand or wrist problems in the last 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
Participants
  No | 109 | 111
  Yes | 7 | 7
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.66, Regression, Logistic; Multiple imputation for missing data was performed. Logistic regression adjusted for sex, age, and duration of symptoms; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.28 to 7.34]

16. Secondary Outcome: Over the Counter Pain Medication 6 Months
Description: Participants were asked if they bought over the counter paracetamol, ibuprofen or co-codamol to help with hand or wrist problems in the last 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
Participants
  No | 82 | 88
  Yes | 34 | 30
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.40, Regression, Logistic; Multiple imputation for missing data was performed. Logistic regression adjusted for sex, age, and duration of symptoms; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.63 to 3.18]

17. Secondary Outcome: Prescribed Pain Medication 6 Months
Description: Participants were asked if they were prescribed tablet medication (paracetamol, ibuprofen, naproxen, diclofenac, codeine, tramadol, co-codomal, tramacet, co-proxamol, dihydrocodeine, other) for hand or wrist problem in the last 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
Participants
  No | 96 | 106
  Yes | 20 | 12
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; The main treatment analyses were based on intention to treat approach; Test type: Superiority; p = 0.20, Regression, Logistic; Multiple imputation for missing data was performed. Logistic regression adjusted for sex, age, and duration of symptoms; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.70 to 5.66]

18. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations Over 24 Months: 6 Weeks
Description: Comparison of overall BCTQ between treatment groups across all time points (6 weeks, 6-, 12-, and 24 month follow-up). Scale 1-5, higher score indicates more severe symptoms and functional impairment. Results are presented at 6 weeks. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 95 | 102
score on a scale | 1.95 (0.82) | 2.30 (0.77)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.001, Mixed Models Analysis — Participants with relevant outcomes reported on at least one follow-up time point were included in the analyses. Adjustment was made for baseline score, age, duration of symptoms, interaction term between treatment and follow-up; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.53 to -0.14]

19. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations Over 24 Months: 6 Months
Description: Comparison of overall BCTQ between treatment groups across all time points (6 weeks, 6-, 12-, and 24 month follow-up. Scale 1-5, higher score indicates more severe symptoms and functional impairment. Results are presented at 6 months. BCTQ: Boston Carpal Tunnel Questionnaire.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 83 | 92
score on a scale | 2.08 (0.79) | 2.04 (0.72)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.74, Mixed Models Analysis — [p-value comment as in outcome 18, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.17 to 0.24]

20. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations Over 24 Months: 12 Months
Description: Comparison of overall BCTQ between treatment groups across all time points (6 weeks, 6-, 12-, and 24 month follow-up). Scale 1-5, higher score indicates more severe symptoms and functional impairment). Results are presented at 12 months. BCTQ: Boston Carpal Tunnel Questionnaire.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 78 | 78
score on a scale | 1.98 (0.88) | 2.05 (0.80)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.41, Mixed Models Analysis — [p-value comment as in outcome 18, analysis 1]; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.30 to 0.12]

21. Secondary Outcome: Secondary: BCTQ Symptom Severity and Functional Limitations Over 24 Months: 24 Months
Description: Comparison of overall BCTQ between treatment groups across all time points (6 weeks, 6-, 12-, and 24 month follow-up). Scale 1-5, higher score indicates more severe symptoms and functional impairment. Results are presented at 24 months. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 70 | 73
score on a scale | 1.79 (0.79) | 1.73 (0.76)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.58, Mixed Models Analysis — [p-value comment as in outcome 18, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.16 to 0.28]

22. Secondary Outcome: Hand-wrist Pain Intensity Over 24 Months: 6 Weeks
Description: Comparison of pain scores between treatment groups across all time points (6 weeks, 6-, 12-, and 24 month follow-up). Scale 0-10, higher score indicates more pain. Results are presented at 6 weeks.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 105 | 106
score on a scale | 3.33 (2.67) | 4.28 (2.62)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.009, Mixed Models Analysis — [p-value comment as in outcome 18, analysis 1]; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-1.72 to -0.24]

23. Secondary Outcome: Hand-wrist Pain Intensity Over 24 Months: 6 Months
Description: Comparison of pain scores between treatment groups across all time points (6 weeks, 6-, 12-, and 24 month follow-up). Scale 0-10, higher score indicates more pain. Results are presented at 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 92 | 94
score on a scale | 4.11 (3.01) | 3.29 (2.74)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.058, Mixed Models Analysis — [p-value comment as in outcome 18, analysis 1]; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-0.02 to 1.54]

24. Secondary Outcome: Hand-wrist Pain Intensity Over 24 Months: 12 Months
Description: Comparison of pain scores between treatment groups across all time points (6 weeks, 6-, 12-, and 24 month follow-up). Scale 0-10, higher score indicates more pain. Results are presented at 12 months.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 83 | 85
score on a scale | 3.17 (2.93) | 3.14 (2.74)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.95, Mixed Models Analysis — [p-value comment as in outcome 18, analysis 1]; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.79 to 0.85]

25. Secondary Outcome: Hand-wrist Pain Intensity Over 24 Months: 24 Months
Description: Comparison of pain scores between treatment groups across all time points (6 weeks, 6-, 12-, and 24 month follow-up). Scale 0-10, higher score indicates more pain. Results are presented at 24 months.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 75 | 77
score on a scale | 2.81 (3.19) | 2.40 (2.83)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.35, Mixed Models Analysis — [p-value comment as in outcome 18, analysis 1]; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-0.45 to 1.26]

26. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Weeks (Complete Case Analysis (CC))
Description: Sensitivity analysis for comparison of overall BCTQ between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms and functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 95 | 102
score on a scale | 1.95 (0.82) | 2.29 (0.77)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p < 0.001, Regression, Linear; Complete case analysis as a sensitivity analysis was performed. Linear regression adjusted for baseline score, sex, age, and duration of symptoms; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.54 to -0.19]

27. Secondary Outcome: BCTQ Symptom Severity Subscale 6 Weeks (CC)
Description: Sensitivity analysis for comparison of BCTQ symptom severity between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms) on participants with complete data. BCTQ:
  Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 104 | 104
score on a scale | 2.07 (0.83) | 2.44 (0.78)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p < 0.001, Regression, Linear; [statistical method as in outcome 26, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.59 to -0.21]

28. Secondary Outcome: BCTQ Functional Limitations Subscale 6 Weeks (CC)
Description: Sensitivity analysis for comparison of overall BCTQ between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 96 | 105
score on a scale | 1.86 (0.91) | 2.10 (0.86)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.005, Regression, Linear; [statistical method as in outcome 26, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.44 to -0.08]

29. Secondary Outcome: Hand-wrist Pain Intensity 6 Weeks (CC)
Description: Sensitivity analysis for comparison of pain scores between treatment groups at 6 weeks follow-up (scale 0-10, higher score indicates more pain) on participants with complete data.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 105 | 106
score on a scale | 3.33 (2.67) | 4.28 (2.62)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.002, Regression, Linear; [statistical method as in outcome 26, analysis 1]; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.72 to -0.38]

30. Secondary Outcome: Insomnia Due to Hand-wrist Problems 6 Weeks (CC)
Description: Participants were asked four questions how hand and wrist problems affects their sleep. Participants reporting hand and wrist problems affects their sleep on most nights on one or more questions were deemed to have insomnia. Sensitivity analysis for comparison of the odds of insomnia between treatment groups at 6 weeks follow-up on participants with complete data.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 97 | 96
Participants
  No | 75 | 62
  Yes | 22 | 34
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.006, Regression, Logistic; Complete case analysis as a sensitivity analysis was performed. Logistic regression adjusted for baseline score, sex, age, and duration of symptoms; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.17 to 0.74]

31. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Months (CC)
Description: Sensitivity analysis for comparison of overall BCTQ between treatment groups at 6 months follow-up (scale 1-5, higher score indicates more severe symptoms and functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 83 | 92
score on a scale | 2.08 (0.79) | 2.04 (0.72)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.58, Regression, Linear; [statistical method as in outcome 26, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.13 to 0.24]

32. Secondary Outcome: BCTQ Symptom Severity Subscale 6 Months (CC)
Description: Sensitivity analysis for comparison of BCTQ symptom severity between treatment groups at 6 months follow-up (scale 1-5, higher score indicates more severe symptoms) on participants with complete data. BCTQ:
  Boston Carpal Tunnel Questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 88 | 94
score on a scale | 2.29 (0.87) | 2.16 (0.74)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.25, Regression, Linear; [statistical method as in outcome 26, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.09 to 0.35]

33. Secondary Outcome: BCTQ Functional Limitations Subscale 6 Months (CC)
Description: Sensitivity analysis for comparison of BCTQ function limitations between treatment groups at 6 months follow-up (scale 1-5, higher score indicates more functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 85 | 93
score on a scale | 1.85 (0.84) | 1.88 (0.82)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.93, Regression, Linear; [statistical method as in outcome 26, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.17 to 0.18]

34. Secondary Outcome: Hand-wrist Pain Intensity 6 Months (CC)
Description: Sensitivity analysis for comparison of pain scores between treatment groups at 6 months follow-up (scale 0-10, higher score indicates more pain) on participants with complete data.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 92 | 94
score on a scale | 4.11 (3.01) | 3.29 (2.74)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.052, Regression, Linear; [statistical method as in outcome 26, analysis 1]; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [-0.01 to 1.61]

35. Secondary Outcome: Insomnia Due to Hand-wrist Problems 6 Months (CC)
Description: Participants were asked four questions how hand and wrist problems affects their sleep. Participants reporting hand and wrist problems affects their sleep on most nights on one or more questions were deemed to have insomnia. Sensitivity analysis for comparison of the odds of insomnia between treatment groups at 6 months follow-up on participants with complete data.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 80 | 86
Participants
  No | 60 | 68
  Yes | 20 | 18
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.53, Regression, Logistic; [statistical method as in outcome 30, analysis 1]; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.58 to 2.88]

36. Secondary Outcome: Referral to Surgery 6 Months (CC)
Description: Participants were asked if they were referred for surgery (carpal tunnel decompression) in the last 6 months. Sensitivity analysis for comparison of the odds of insomnia between treatment groups at 6 months follow-up on participants with complete data.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 96 | 93
Participants
  No | 80 | 82
  Yes | 16 | 11
Statistical Analysis 1: Comparison: Steroid Injection; Test type: Superiority; p = 0.41, Regression, Logistic; Complete case analysis as a sensitivity analysis was performed. Logistic regression adjusted for sex, age, and duration of symptoms; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.61 to 3.34]

37. Secondary Outcome: Herbal Remedies and Vitamin Use 6 Months (CC)
Description: Participants were asked if they had bought herbal remedies or vitamins to help with hand or wrist problems in the last 6 months. Sensitivity analysis for comparison of the odds of herbal remedies and vitamin use between treatment groups at 6 months follow-up on participants with complete data.
  Complete case analysis as a sensitivity analysis was planned. Comparison of outcome between treatment arms planned to adjust for sex, age, and duration of symptoms. Logistic regression was not performed due to small number of 'yes' counts.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 80 | 83
Participants
  No | 78 | 81
  Yes | 2 | 2

38. Secondary Outcome: Over the Counter Pain Medication 6 Months (CC)
Description: Participants were asked if they bought over the counter paracetamol, ibuprofen or co-codamol to help with hand or wrist problems in the last 6 months. Sensitivity analysis for comparison of the odds of medication use between treatment groups at 6 months follow-up on participants with complete data.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 80 | 83
Participants
  No | 64 | 66
  Yes | 16 | 17
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.52, Regression, Logistic; [statistical method as in outcome 36, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.57 to 3.06]

39. Secondary Outcome: Prescribed Pain Medication 6 Months (CC)
Description: Participants were asked if they were prescribed tablet medication (paracetamol, ibuprofen, naproxen, diclofenac, codeine, tramadol, co-codomal, tramacet, co-proxamol, dihydrocodeine, other) for hand or wrist problem in the last 6 months. Sensitivity analysis for comparison of the odds of pain medication use between treatment groups at 6 months follow-up on participants with complete data.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 82 | 86
Participants
  No | 70 | 79
  Yes | 12 | 7
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.18, Regression, Logistic; [statistical method as in outcome 36, analysis 1]; Odds Ratio (OR) = 2.05, 95% CI 2-sided [0.72 to 5.78]

40. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Weeks (Per-Protocol Analysis (PP))
Description: Per protocol analysis for comparison of overall BCTQ between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms and functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 94 | 85
score on a scale | 1.96 (0.84) | 2.28 (0.72)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p < 0.001, Regression, Linear; Per protocol analysis on complete date was performed. Linear regression adjusted for baseline score, sex, age, and duration of symptoms; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.55 to -0.18]

41. Secondary Outcome: BCTQ Symptom Severity Subscale 6 Weeks (PP)
Description: Per protocol analysis for comparison of BCTQ symptom severity between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms) on participants with complete data. BCTQ:
  Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 102 | 86
score on a scale | 2.07 (0.83) | 2.44 (0.74)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p < 0.001, Regression, Linear; [statistical method as in outcome 40, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.59 to -0.19]

42. Secondary Outcome: BCTQ Functional Limitations Subscale 6 Weeks (PP)
Description: Per protocol analysis for comparison of BCTQ functional limitations between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more functional impairment) on participants with complete data.
  BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 95 | 87
score on a scale | 1.88 (0.94) | 2.06 (0.80)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.003, Regression, Linear; [statistical method as in outcome 40, analysis 1]; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.46 to -0.09]

43. Secondary Outcome: Hand-wrist Pain Intensity 6 Weeks (PP)
Description: Per protocol analysis for comparison of pain scores between treatment groups at 6 weeks follow-up (higher score indicates more pain) on participants with complete data.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 103 | 87
score on a scale | 3.33 (2.67) | 4.44 (2.50)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.001, Regression, Linear; [statistical method as in outcome 40, analysis 1]; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-1.85 to -0.48]

44. Secondary Outcome: Insomnia Due to Hand-wrist Problems 6 Weeks (PP)
Description: Participants were asked four questions how hand and wrist problems affects their sleep. Participants reporting hand and wrist problems affects their sleep on most nights on one or more questions were deemed to have insomnia. Per protocol analysis for comparison of the odds of insomnia between treatment groups at 6 weeks follow-up on participants with complete data.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 95 | 87
Participants
  No | 74 | 57
  Yes | 21 | 30
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.007, Regression, Logistic; Per protocol analysis on complete date was performed. Logistic regression adjusted for baseline score, sex, age, and duration of symptoms; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.16 to 0.74]

45. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Months (PP)
Description: Per protocol analysis for comparison of overall BCTQ between treatment groups at 6 months follow-up (scale 1-5, higher score indicates more severe symptoms and functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 83 | 76
score on a scale | 2.09 (0.79) | 2.02 (0.69)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.63, Regression, Linear; [statistical method as in outcome 40, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.15 to 0.25]

46. Secondary Outcome: BCTQ Symptom Severity Subscale 6 Months (PP)
Description: Per protocol analysis for comparison of BCTQ symptom severity between treatment groups at 6 months follow-up (scale 1-5, higher score indicates more severe symptoms) on participants with complete data. BCTQ:
  Boston Carpal Tunnel Questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 88 | 78
score on a scale | 2.28 (0.86) | 2.15 (0.73)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.28, Regression, Linear; [statistical method as in outcome 40, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.10 to 0.35]

47. Secondary Outcome: BCTQ Functional Limitations Subscale 6 Months (PP)
Description: Per protocol analysis for comparison of BCTQ functional limitations between treatment groups at 6 months follow-up (scale 1-5, higher score indicates more functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 85 | 77
score on a scale | 1.89 (0.87) | 1.84 (0.77)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.900, Regression, Linear; [statistical method as in outcome 40, analysis 1]; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.18 to 0.20]

48. Secondary Outcome: Hand-wrist Pain Intensity 6 Months (PP)
Description: Per protocol analysis for comparison of pain scores between treatment groups at 6 months follow-up (scale 0-10, higher score indicates more pain) on participants with complete data.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 92 | 78
score on a scale | 4.11 (2.99) | 3.38 (2.79)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.09, Regression, Linear; [statistical method as in outcome 40, analysis 1]; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-0.11 to 1.59]

49. Secondary Outcome: Insomnia Due to Hand-wrist Problems 6 Months (PP)
Description: Participants were asked four questions how hand and wrist problems affects their sleep. Participants reporting hand and wrist problems affects their sleep on most nights on one or more questions were deemed to have insomnia. Per protocol analysis for comparison of the odds of insomnia between treatment groups at 6 months follow-up on participants with complete data.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 81 | 75
Participants
  No | 61 | 59
  Yes | 20 | 16
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.58, Regression, Logistic; [statistical method as in outcome 44, analysis 1]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.56 to 2.85]

50. Secondary Outcome: Referral to Surgery at 6 Months (PP)
Description: Participants were asked if they were referred for surgery (carpal tunnel decompression) in the last 6 months. Per protocol analysis for comparison of the odds of surgery between treatment groups at 6 months follow-up on participants with complete data.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 94 | 85
Participants
  No | 78 | 74
  Yes | 16 | 11
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.52, Regression, Logistic; Per protocol analysis on complete date was performed. Logistic regression adjusted for sex, age, and duration of symptoms; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.57 to 3.01]

51. Secondary Outcome: Herbal Remedies and Vitamin Use 6 Months (PP)
Description: Participants were asked if they had bought herbal remedies or vitamins to help with hand or wrist problems in the last 6 months. Per protocol analysis for comparison of the odds of herbal remedies and vitamin use between treatment groups at 6 months follow-up on participants with complete data.
  Per protocol analysis on complete date was planned. Comparison of outcome between treatment arms planned to adjust for sex, age, and duration of symptoms. Logistic regression was not performed due to small number of 'yes' counts.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 81 | 73
Participants
  No | 78 | 72
  Yes | 3 | 1

52. Secondary Outcome: Over the Counter Pain Medication 6 Months (PP)
Description: Participants were asked if they bought over the counter paracetamol, ibuprofen or co-codamol to help with hand or wrist problems in the last 6 months. Per protocol analysis for comparison of the odds of medication use between treatment groups at 6 months follow-up on participants with complete data
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 81 | 73
Participants
  No | 65 | 58
  Yes | 16 | 15
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.61, Regression, Logistic; [statistical method as in outcome 50, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.53 to 2.95]

53. Secondary Outcome: Prescribed Pain Medication 6 Months (PP)
Description: Participants were asked if they were prescribed tablet medication (paracetamol, ibuprofen, naproxen, diclofenac, codeine, tramadol, co-codomal, tramacet, co-proxamol, dihydrocodeine, other) for hand or wrist problem in the last 6 months. Per protocol analysis for comparison of the odds of medication use between treatment groups at 6 months follow-up on participants with complete data.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 83 | 76
Participants
  No | 70 | 70
  Yes | 13 | 6
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.14, Regression, Logistic; [statistical method as in outcome 50, analysis 1]; Odds Ratio (OR) = 2.24, 95% CI 2-sided [0.77 to 6.58]

54. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Weeks (Subgroup Analysis (SG), Intervention of Their Preference)
Description: Subgroup analysis was performed in patients who were allocated the intervention of their preference. Comparison of overall BCTQ between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms and functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 24 | 18
score on a scale | 1.88 (0.76) | 2.19 (0.75)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.014, Regression, Linear; Sub group analysis on complete data was performed. Linear regression adjusted for baseline score, sex, age, and duration of symptoms; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.93 to -0.12]

55. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Weeks (SG, Did Not Receive the Intervention of Their Preference)
Description: Subgroup analysis was performed in patients who did not receive the intervention of their preference. Comparison of overall BCTQ between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms and functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 18 | 34
score on a scale | 2.15 (0.91) | 2.40 (0.84)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.53, Regression, Linear; [statistical method as in outcome 54, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.50 to 0.26]

56. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Weeks (SG, Did Not State a Preference of Intervention)
Description: Subgroup analysis was performed in patients who did not state a preference of intervention. Comparison of overall BCTQ between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms and functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 67 | 61
score on a scale | 2.03 (0.79) | 2.26 (0.69)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.015, Regression, Linear; [statistical method as in outcome 54, analysis 1]; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.44 to -0.05]

57. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Weeks (SG, Preferred Injection)
Description: Subgroup analysis was performed in patients who preferred injection. Comparison of overall BCTQ between treatment groups at 6 weeks follow-up (scale 1-5, higher score indicates more severe symptoms and functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 24 | 34
score on a scale | 1.88 (0.76) | 2.40 (0.84)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.002, Regression, Linear; [statistical method as in outcome 54, analysis 1]; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-0.97 to -0.23]

58. Secondary Outcome: BCTQ Symptom Severity and Functional Limitations 6 Weeks (SG, Preferred Splint)
Description: Subgroup analysis was performed in patients who preferred splint. Comparison of overall BCTQ between treatment groups at 6 weeks follow-up (higher score indicates more severe symptoms and functional impairment) on participants with complete data. BCTQ: Boston Carpal Tunnel Questionnaire
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 18 | 34
score on a scale | 2.15 (0.91) | 2.40 (0.84)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; p = 0.25, Regression, Linear; [statistical method as in outcome 54, analysis 1]; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.60 to 0.16]

59. Secondary Outcome: NHS Cost Differences at 6 Months
Description: Cost of interventions at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: UK Pounds
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
UK Pounds | 346.78 (467.97) | 313.24 (480.84)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; Regression, Linear; Comparison of outcome between treatment groups performed on multiply imputed data; Mean Difference (Final Values) = 33.54, 95% CI 2-sided [-94.57 to 145.59]

60. Secondary Outcome: NHS Cost Differences at 6 Months (CC)
Description: Complete case analysis on the cost of interventions at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: UK Pounds
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
UK Pounds | 353.48 (512.85) | 306.42 (524.51)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; Regression, Linear; Comparison of outcome between treatment groups on complete data; Mean Difference (Final Values) = 47.06, 95% CI 2-sided [-104.84 to 187.31]

61. Secondary Outcome: NHS Cost Differences at 12 Months
Description: Cost of interventions at 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: UK Pounds
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
UK Pounds | 508.69 (657.48) | 395.54 (596.47)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; Regression, Linear; Comparison of outcome between treatment groups; Mean Difference (Final Values) = 113.15, 95% CI 2-sided [-37.09 to 279.21]

62. Secondary Outcome: NHS Cost Differences at 24 Months
Description: Cost of interventions at 24 months
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: UK Pounds
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
UK Pounds | 657.87 (808.57) | 586.77 (783.45)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; Regression, Linear; Comparison of outcome between treatment groups; Mean Difference (Final Values) = 71.1, 95% CI 2-sided [-120.84 to 291.24]

63. Secondary Outcome: QALYS at 6 Months (Cross-walk Tariff)
Description: The Quality Adjusted Life Years (QALYs) is a measure of the state of health of a person/group in which the benefits, in terms of length of life, are adjusted to reflect the quality of life. One QALY is equal to 1 year of life in perfect health. QALYs are calculated by estimating the years of life remaining for a patient following a particular treatment/intervention and weighting each year with a quality-of-life score (on a 0 to 1 scale). It is often measured in terms of the person's ability to carry out the activities of daily life and freedom from pain and mental disturbance. The QALY does not have a maximum score.
  Cross-walk tariff: Crosswalk value sets were developed from a study of respondents who completed both the EQ-5D-3L and EQ-5D-5L. The crosswalk used a non-parametric response mapping method to predict values that are linked to the EQ-5D-3L value set. In short, the cross-walk tariff maps EQ-5D-5L values.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
score on a scale | 0.354 (0.093) | 0.356 (0.087)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.01 to 0.02]

64. Secondary Outcome: QALYS at 12 Months (Cross-walk Tariff)
Description: as for outcome 63
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
score on a scale | 0.723 (0.163) | 0.736 (0.156)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.034 to 0.027]

65. Secondary Outcome: QALYS at 24 Months (Cross-walk Tariff)
Description: as for outcome 63
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Steroid Injection | Wrist Splint
Number analyzed (Participants) | 116 | 118
score on a scale | 1.461 (0.311) | 1.497 (0.301)
Statistical Analysis 1: Comparison: Steroid Injection vs Wrist Splint; Test type: Superiority; Regression, Linear; Mean Difference (Final Values) = -0.022, 95% CI 2-sided [-0.093 to 0.045]

ADVERSE EVENTS:
Time Frame: 24 months
Description: Reporting by investigators. Expected related adverse events self-reported by participants in 6-week questionnaire.
Arm/Group | Steroid Injection | Wrist Splint
All-Cause Mortality (participants affected / at risk) | 2/116 | 0/118
Serious Adverse Events (participants affected / at risk) | 3/116 | 4/118
Other Adverse Events (participants affected / at risk) | 57/116 | 7/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroid Injection (N=116) | Wrist Splint (N=118)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Open comminuted fracture left middle finger, operative fixation with K-wires
Other (Cardiac disorders) | 1 (1) | 0 (0) — Cardiac failure NB No specific adverse event term for this AE in CTCAE 4.0. Adverse event recorded as 'other' & AE Term Additional Description provided, aligning with trial EudraCT entry.
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cryptogenic organising pneumonia NB No specific adverse event term for this AE in CTCAE 4.0. Adverse event recorded as 'other' & AE Term Additional Description provided, aligning with trial EudraCT entry.
Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patella resurfacing NB No specific adverse event term for this AE in CTCAE 4.0. Adverse event recorded as 'other' & AE Term Additional Description provided, aligning with trial EudraCT entry.
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Total arthroplasty for osteoarthritis (one hip, one knee)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroid Injection (N=116) | Wrist Splint (N=118)
Flushing (Vascular disorders) | 17 (17) | 0 (0)
Other (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) — Thinning, lightening or darkening of skin at injection site
Arthralgia (Musculoskeletal and connective tissue disorders) | 53 (53) | 7 (7) — For steroid injection, hand or wrist was more painful following injection. For splinting, participants unable to wear splint because of discomfort.

LIMITATIONS AND CAVEATS:
Trial participants and clinicians were not masked to treatment allocation. We recruited six short of the target 240 participants; however, statistical power was retained because of higher than anticipated follow-up rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No